CLINICAL TRIAL: NCT04298411
Title: Project Falcon: Exploring a Virtual Reality-based Video Game With Haptic Feedback for Sensory-motor Rehabilitation of Young People With Cerebral Palsy
Brief Title: Project Falcon: Exploring a Virtual Reality-based Video Game for Young People With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-530
Record Dates: First submitted 2020-01-29; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Palsy
Keywords: haptic feedback; Novint Falcon; upper limb motor function; rehabilitation; motor learning; neuroplasticity; video games
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Participants will take part in 12 one-hour rehabilitation sessions over 12 weeks in the clinic at Holland Bloorview Kids Rehabilitation Hospital and Institut de réadaptation en déficience physique de Québec, during which they will play games developed for the Novint Falcon.
  Interventions: Device: Falcon

INTERVENTIONS:
Device: Falcon — The Falcon contains a selection of 25+ games that require wrist extension and challenges children to grasp the controller with their affected hand. As children progress, they may advance to more difficult games that challenge the child to work against a resistance and/or apply greater grip forces. Therapists will be trained on the system, games, and given a guide summarizing the available games and the motor function areas targeted in the game. Using this guide, therapists can choose the games that are most suited to the child's abilities and goals. As multiple games will target many of the same motor function areas, children will have the option of choosing the games they like best to maximize motivational value. While this introduces some variability in the intervention, this flexibility is required to ensure that the therapy is targeting the specific interests, needs and goals of each individual child and is reflective of how ICP is used in a clinic setting.

SUMMARY:
This study seeks to 1) adapt a low-cost controller, the Novint Falcon, and a set of video games that would provide rehabilitative feedback for young people with cerebral palsy, and 2) explore feasibility of the Falcon system and it's effect on upper limb and hand function.

DETAILED DESCRIPTION:
Motivation: Children with cerebral palsy (CP) experience various challenges in upper limb motor function (e.g. muscle weakness, impaired manual abilities, spasticity, ataxia, athetosis and/or dystonia) that can impede their activities and participation in daily life. Rehabilitation strategies to support children with CP in achieving improved upper limb control target these areas through strengthening, endurance building, and motor learning activities. Neuroplasticity and motor learning are promoted by repetitive practice in a motivating and rewarding environment, immediate feedback on performance, and use of tasks with appropriate complexity that is increased as progress is made. Many elements of video games (e.g. progressive difficulty levels, engaging game play) may support motor learning and early evidence suggests that interactive computer play is likely effective for improving lower limb function with some promising indications for upper limb rehabilitation. The majority of evidence comes from studies that have used commercial gaming systems where children interact with virtual objects on the screen via their movements. These systems, however, do not provide haptic feedback, which may aid in motor learning and the transference of skills practiced in virtual environments to real-life.

The Novint Falcon is a low-cost, three degree-of-freedom video game controller that can provide force and tactile feedback during game play. The three motors that enable the provision of haptic feedback can also be used to assist movements. A software development kit is available and enables custom design of games and applications. One previous study investigated this device in adults for stroke rehabilitation. While promising, one drawback identified was that the available mini-games did not practice therapeutically relevant movements.

Objective: Considering the upper limb motor challenges experienced by children with CP and the potential of the Novint Falcon to assist in their rehabilitation, research is needed to develop challenging video games adapted for this controller. The objectives of this proposal are 1) to adapt a low-cost haptic controller and compile a set of video games that provide tactile and force feedback for the rehabilitation of young people with CP, and 2) to explore the feasibility of the system and the effects on upper limb and hand function.

Methods: In pursuit of these two objectives:

1. Existing mini-games will be reviewed in partnership with therapists to identify promising games. Thereafter, new mini-games will be designed as needed to meet with therapeutic goals identified by the therapists. The design of the controller's grip will then be reviewed via a participatory design approach that engages both therapists and children with CP. New grips will be created as needed.
2. The resulting system will be evaluated in a clinic setting by children with hemiplegic CP (ages 7 to 16 years; n=14; 7/site) at Holland Bloorview Kids Rehabilitation Hospital and Institut de réadaptation en déficience physique de Québec. Each child with CP will take part in one initial assessment session, 12 one-hour rehabilitation sessions over 12 weeks during which they will play games developed for the Novint Falcon, and one final assessment session. Independent evaluators will assess the children with CP before (two baseline measurements will be established) and after the 12-week intervention. The outcomes of interest include: Canadian Occupational Therapy Performance Measure, Quality of Upper Extremity Skills Test, sensory profile, grip strength, and upper extremity range of motion. Further, child participants will complete the Physical Activity Enjoyment Scale, while therapists will complete the System Usability scale.

Expected Outcomes. The results of this study if promising, will lay the foundation for a CIHR grant to explore the role of haptic feedback in interactive computer play therapies. Through this research, the investigators hope to offer an appealing tool to aid in the rehabilitation of children with CP that is both therapeutically valuable and enjoyable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegic cerebral palsy
* Level I to III on the Manual Abilities Classification System (MACS)
* Ability to understand and communicate in English (Holland Bloorview site) or French (IRDPQ site) at a grade 2 level or higher

Exclusion Criteria:

* Received Botulinum Toxin in the most recent 3 months
* History of epilepsy
* Past experience of an injury or disability that would render therapy unsafe
* Visual, cognitive or auditory disabilities that interfere with the ICP

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) | Measured at 0 weeks (pre-intervention) and 12 weeks (post-intervention).
  The Canadian Occupational Performance Measure evaluates changes in perceived function and satisfaction of performance in self-identified goal areas. The child and parent work together with the therapist to identify 1-3 goals of interest. For each goal area, the child/parent ranks its importance, performance and satisfaction on a scale of 1-10. A higher rating indicates a more positive outcome.

SECONDARY OUTCOMES:
Change in Grip Strength | Measured at 0 weeks (pre-intervention) and 12 weeks (post-intervention).
  A sphygmomanometer is used to measure grip strength of the hand by determining the amount of pressure (mmHg) that the hand can apply.
active/passive range of motion | Measured at 0 weeks (pre-intervention) and 12 weeks (post-intervention).
  A goniometer is used to measure degrees of active/passive range of motion of the wrist.
Change in Children's Hand-use Experience Questionnaire (CHEQ) | Measured at 0 weeks (pre-intervention) and 12 weeks (post-intervention).
  Children's Hand-use Experience Questionnaire (CHEQ) is a 29 item child- or parent- completed questionnaire that examines how the weaker/affected limb is used in everyday activities. It presents a list of common daily activities that typically require use of two hands.The minimum score value is 0 and the maximum score value is 100. A higher score means a better outcome.
Change in Shortened Physical Activity Enjoyment Scale (S-PACES) | Measured at 1 week, 6 weeks, and 12 weeks.
  Consists of 10 pairs of statements scored on a 5-point Likert scale that probe factors in enjoyment of physical activity. The minimum score value is 1 and the maximum score value is 5. A higher score means a better outcome.
Change in the answers reported in custom feedback questionnaires | Measured at 1 week, 6 weeks, and 12 weeks.
  Custom feedback questionnaires will be used to evaluate the perceived quality of feedback, motivation, and difficulty of tasks during ICP therapies. It is based on validated questionnaires for measuring usability (SUS) and enjoyment (Flow short) and a custom questionnaire used in a previous study investigating ICP therapy games with this population. The custom feedback questionnaire consists of open-ended questions.
  Open-ended questions include: What did you like about the games? What didn't you like about the games? What would make the games more fun?

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Holland Bloorview Kid's Rehabilitation Hospital; Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Centre interdisciplinaire de recherche en réadaptation et en intégration sociale, Québec

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plans.